CLINICAL TRIAL: NCT04049500
Title: An Observational Study to Adapt a Digital Diabetes Prevention Program (dDPP) and Incorporate it Into the Clinical Workflows.
Brief Title: Adapt and Incorporate dDPP Into Clinical Workflows
Status: Withdrawn | Type: Observational
Why Stopped: study was never started
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-00758
Record Dates: First submitted 2019-08-01; First posted 2019-08-08 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Physician-Patient Relations; Nurse-Patient Relations
Keywords: Physicians; Nurses; Practice assistants; Health coaches; Population health managers; Patient navigators

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinicians: Five practices will be selected from NYULH ambulatory practice sites to represent the spectrum of provider settings within the system. These sites will be the clinical partners for the adaptation of the dDPP tool suite
  Interventions: Other: Digital Diabetes Prevention Program (dDPP)

INTERVENTIONS:
Other: Digital Diabetes Prevention Program (dDPP) — dDPP tool suite to integrate with the EHR and clinical workflows

SUMMARY:
This observational study will seek to adapt a digital diabetes prevention program (dDPP) tool suite into clinical workflows. This tool pushes key dDPP data elements (e.g. weight and daily step count) directly into EHR workflows of primary care to enhance patient engagement. It seeks to determine the impact of combining adapted visualizations and summaries of key dDPP data elements directly into the EHR with automated notifications and messaging designed to enhance patient engagement in the dDPP. The study will involve provider workflow analysis based on observation and facilitated group tool adaptation sessions.

DETAILED DESCRIPTION:
Primary objective: to examine the impact of the dDPP tool suite on the EHR and clinical workflows, and identify optimization opportunities.

Secondary objective: to assess the "usability" of the proposed dDPP tool suite in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Physicians
* Nurses
* Practice assistants
* Health coaches
* Population health managers
* Patient navigators

Exclusion Criteria:

* Practices will be ineligible for participation if they treat fewer than 100 adults with prediabetes.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Five practices will be selected from NYULH ambulatory practice sites to represent the spectrum of provider settings within the system. These sites will be the clinical partners for the adaptation of the dDPP tool suite.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Usability will be assessed using a 5-point Likert scale | 12 Months
  5 point likert scale is measured on a 5 point scale, 1 being "very unsatisfied" and 5 being "very satisfied." Higher scores mean more usability

CONTACTS AND LOCATIONS:
Overall Officials: Devin Mann, MD, Principal Investigator — NYU Langone

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).Upon reasonable request.Requests should be directed to devin.mann@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.

REFERENCES:
- [Derived] Rodriguez DV, Lawrence K, Gonzalez J, Brandfield-Harvey B, Xu L, Tasneem S, Levine DL, Mann D. Leveraging Generative AI Tools to Support the Development of Digital Solutions in Health Care Research: Case Study. JMIR Hum Factors. 2024 Mar 6;11:e52885. doi: 10.2196/52885. PMID 38446539
- [Derived] Lawrence K, Rodriguez DV, Feldthouse DM, Shelley D, Yu JL, Belli HM, Gonzalez J, Tasneem S, Fontaine J, Groom LL, Luu S, Wu Y, McTigue KM, Rockette-Wagner B, Mann DM. Effectiveness of an Integrated Engagement Support System to Facilitate Patient Use of Digital Diabetes Prevention Programs: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Feb 9;10(2):e26750. doi: 10.2196/26750. PMID 33560240